CLINICAL TRIAL: NCT03278275
Title: PET/CT Imaging of uPAR-expression in Patients With Neuroendocrine Tumors Using 68Ga-NOTA-AE105
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Esben Carlsen, Principle investigator, Medical doctor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK2017-1; 2017-002312-13 (EudraCT Number)
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Neuroendocrine Tumors
Keywords: urokinase plasminogen activator receptor; uPAR PET/CT; positron emission tomography; neuroendocrine tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- uPAR PET/CT (Experimental): One injection of the radioligand 68Ga-NOTA-AE105
  Interventions: Drug: One injection of 68Ga-NOTA-AE105; Device: PET/CT

INTERVENTIONS:
Drug: One injection of 68Ga-NOTA-AE105 — One injection of 68Ga-NORA-AE105
Device: PET/CT — Following injection of 68Ga-NOTA-AE105 the participants will be subjected to whole body PET/CT

SUMMARY:
The aim of this non-randomised, prospective study is to investigate the applicability and prognostic value of uPAR PET/CT with the radioligand 68Ga-NOTA-AE105 in patients with neuroendocrine tumors (NETs).

DETAILED DESCRIPTION:
68Ga-NOTA-AE105 is a radioligand targeting urokinase plasminogen activator receptor (uPAR), which is a promising imaging biomarker of tumor aggressiveness. A total of 120 NET patients will be subjected to a uPAR-PET/CT scan. Follow-up will be performed (from the time of the angiogenesis PET/ CT) at 6 months for disease specific survival (DSS) and a 1 year follow-up for PFS and OS. The uptake of 68Ga-NOTA-AE105 in tumor lesions will be quantified as Standardized Uptake Values (SUVmax/SUVmean) and compared with PFS, DSS and OS (dichotomized above/below median SUVmax and analyzed by Kaplan-Meier)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gastro-entero-pancreatic Neuroendocrine Tumors (GEP-NET; grade: G1-G3) or broncho-pulmonary NET.
* WHO performance status 0-2
* Must be able to read and understand the patient information in Danish and to give informed consent

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Weight more than the maximum weight limit for the PET/CT bed of the scanner (140 kg)
* History of allergic reaction attributable to compounds of similar chemical or biologic composition to 68Ga-NODAGA-E[c(RGDyK)]2
* In case of broncho-pulmonary NET, the subtype must not be small cell lung cancer (SCLC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
uPAR PET/CT imaging of patients with neuroendocrine tumors | 1 hour
  The radioligand 68Ga-NOTA-AE105 can be used to visualize neuroendocrine tumors (grade G1-G3)

SECONDARY OUTCOMES:
uPAR PET/CT prognostic factor for progression free survival | 12 months
  The uptake of the 68Ga-NOTA-AE105 in neuroendocrine tumor lesions (quantified as Standard Uptake Values) is associated with progression free survival (PFS) neuroendocrine tumors (grade G1-G3)
uPAR PET/CT prognostic factor for overall and disease specific survival | 12 months
  The uptake of the 68Ga-NOTA-AE105 in neuroendocrine tumor lesions (quantified as Standard Uptake Values) is associated with overall and disease specific free survival (PFS) neuroendocrine tumors (grade G1-G3)

CONTACTS AND LOCATIONS:
Overall Officials: Esben Carlsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Denmark